CLINICAL TRIAL: NCT01651637
Title: A First in Human Clinical Study on the Safety and Tolerability of Two Escalating Single Doses of CHF 5633 (Synthetic Surfactant) in Preterm Neonates With Respiratory Distress Syndrome
Brief Title: First In Human Study on Synthetic Surfactant CHF 5633 in Respiratory Distress Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCD-1011-PR-0059
Record Dates: First submitted 2012-04-20; First posted 2012-07-27 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Respiratory Distress Syndrome in Premature Infants
Keywords: Respiratory Distress syndrome; Complications of prematurity
MeSH Terms: conditions — Respiratory Distress Syndrome In Premature Infants; Respiratory Distress Syndrome | interventions — Surface-Active Agents; CHF5633

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Synthetic Surfactant (Experimental): Cohort Design
  Interventions: Drug: synthetic surfactant (CHF5633)

INTERVENTIONS:
Drug: synthetic surfactant (CHF5633) — CHF5633 100 mg/kg; CHF5633 200 mg/kg synthetic surfactant sterile suspension in 3.0 ml glass vials with a total concentration of 80 mg/ml for intratracheal administration. Single administration

SUMMARY:
The aim of this study is to investigate the safety and tolerability of intratracheal administration of two different single doses of CHF 5633 in preterm neonates with RDS in terms of adverse events, adverse drug reactions, hematology and biochemistry values, the incidence of major neonatal morbidities including bronchopulmonary dysplasia (BPD) and mortality.

DETAILED DESCRIPTION:
The study will be a multicentre, open-label, single escalating dose, per-cohort design.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained by parents/legal representative (according to local regulation) prior to any study-related procedures
* Inborn and outborn, preterm neonates of either sex with a gestational age of 27 weeks up to 33 weeks+6
* Clinical and radiological findings typical of RDS
* Age on admission to the study < 24 hours from birth
* Requirement of endotracheal intubation for surfactant administration
* Fraction of inspired oxygen (FiO2) > 0.35 to maintain SpO2 between 90-95 %
* Documentation of normal cranial ultrasound scan

Exclusion Criteria:

* Use of surfactant prior to study entry and need for intratracheal administration of any other treatment (e.g. nitric oxide)
* Known genetic or chromosomal disorders, major congenital anomalies (cardiac malformations, myelomeningocele etc)
* Maternal drug abuse (heroin, methadone, methamphetamine, or cocaine) or significant alcohol consumption during pregnancy
* Clinical chorioamnionitis (Appendix III)
* Strong suspicion of congenital pneumonia/infection, sepsis
* Evidence of severe birth asphyxia or a 5 minutes Apgar score less / equal 3
* Presence of air leaks prior to study entry
* Neonatal seizures prior to study entry
* Mothers with prolonged rupture of the membranes (> 3 weeks duration)
* Any condition that, in the opinion of the Investigator, would place the neonate at undue risk
* Participation in another clinical trial of any placebo, drug or biological substance conducted under the provisions of a protocol

Ages: 27 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2015-01-23 (Actual); Study Completion 2015-01-23 (Actual)

PRIMARY OUTCOMES:
Monitoring of adverse events following CHF5633 administration | For duration of hospital stay (expected average of 9 weeks)

SECONDARY OUTCOMES:
CHF 5633 efficacy profile (oxygenation , ventilatory requirements and need for rescue surfactant treatment),systemic absorption and immunogenicity assesment | At min 30, at hrs 1, 3, 6, 12, 24, at days 2, 3, 7 and at days 10, 28, at 36 weeks pma post dosing for ventilatory requirements, at pre-dose and 3 hrs and 24 hrs post dosing for systemic absorption and at 8 wks after administration for immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Christian Speer, MD, Principal Investigator — Universitäts-Kinderklinik Würzburg (Germany)
Locations (1):
- Liverpool Women's Hospital Neonatal Unit Liverpool Women's Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sweet DG, Turner MA, Stranak Z, Plavka R, Clarke P, Stenson BJ, Singer D, Goelz R, Fabbri L, Varoli G, Piccinno A, Santoro D, Speer CP. A first-in-human clinical study of a new SP-B and SP-C enriched synthetic surfactant (CHF5633) in preterm babies with respiratory distress syndrome. Arch Dis Child Fetal Neonatal Ed. 2017 Nov;102(6):F497-F503. doi: 10.1136/archdischild-2017-312722. Epub 2017 May 2. PMID 28465315
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2011-001331-22